CLINICAL TRIAL: NCT06958406
Title: Lesion-Network Mapping Analysis With Brain Connectomics to Reveal the Neural Mechanisms of Cerebrocardiac Syndrome Following Traumatic Brain Injury
Brief Title: Neural Mechanism of Cerebrocardiac Syndrome Following Traumatic Brain Injury
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Hao Chen, MD, PhD, Associate Professor, Chief Physician, Graduate Supervisor, Shanghai 6th People's Hospital
Other Study IDs: 2024-KY-136（K）
Record Dates: First submitted 2025-03-03; First posted 2025-05-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Traumatic Brain Injury; Cerebrocardiac Syndrome
Keywords: traumatic brain injury; cerebrocardiac syndrome; brain connectomics
MeSH Terms: conditions — Brain Injuries, Traumatic; Neurocirculatory Asthenia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- TBI-CCS: Patients with TBI-induced CCS, including myocardial injury, arrhythmia or heart failure.
- Non TBI-CCS: Patients with non TBI-induced CCS.
- Normal control: Normal healthy people.

SUMMARY:
Cerebrocardiac syndrome (CCS), including myocardial injury, arrhythmia or heart failure is one of serious complications of traumatic brain injury (TBI), mostly occurs within seven days after TBI, which directly aggravates the brain damage and affects the prognosis of TBI patients. Accumulative evidences suggest that autonomic nervous system disorder is a key initiation point for CCS, but how TBI affects the specific action patterns is not yet clear. Therefore, elucidating the neural mechanisms of TBI-induced CCS, maintaining the central sympathetic-parasympathetic balance through novel interventions such as noninvasive brain stimulation, may fundamentally block the downstream peripheral mechanism, thus achieving effective prevention and treatment for CCS. Based on the current emerging research in brain connectomics and lesion-symptom mapping, we speculate that cerebral contusions can cause structural or functional disconnection of key nodes in the central autonomic nervous system regulatory network, thereby mediating the occurrence of TBI-induced CCS.

In this study, magnetic resonance imaging (MRI) or functional MRI (fMRI) examinations were performed in patients with mild or moderate TBI with aim to explore the association between structural and functional disconnection caused by cerebral contusion and TBI-induced CCS, and to screen out the neural anatomical structures to predict CCS following TBI, providing therapy targets for prevention and treatment of CCS.

ELIGIBILITY:
Inclusion Criteria:

* Patients with isolated closed head trauma
* Age 18-80 years old
* Admitted to hospital within 24 hours of injury
* Mild or moderate TBI (Glasgow Coma Scale score of 9-15)
* Signed consent form

Exclusion Criteria:

* Severe TBI (Glasgow Coma Scale score of 3-8)
* A history of stroke, TBI, intracranial tumor or surgery in the past 1 year
* A history of coronary heart disease, structural heart disease and other primary heart diseases or suspected cardiac symptoms prior to injury
* Causes of abnormal cardiac biomarkers such as renal insufficiency, severe anemia, sepsis, cardiotoxic drugs and so on
* Not suitable for MRI examinations, such as pregnant women and those with metal implants in the body
* Undergo surgery prior to MRI examinations or cardiac testing

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Traumatic brain injury patients and healthy volunteers.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05-06 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Brain network evaluation by MRI | Within 3 days after enrollment
  MRI data of all participants are acquired within 3 days after enrollment, and the MRI scans include one or more of the following contents：
  1. 3D T1-weighted images, which were acquired with a magnetization prepared rapid-acquisition gradient-echo sequence.
  2. The resting state-fMRI data, acquired with an interleaved T2-weighted axial gradient-echo echoplanar imaging sequence.
  3. DTI datasets, acquired using a fully-sampled spin-echo EPI sequence.
Cardiac evaluation by ECG | Within 3 days after enrollment
  ECG data of all participants are acquired within 3 days after enrollment, and include resting and ambulatory ECG to detect arrhythmias, heart rate variability or myocardial ischemia. Specifically, arrhythmias include atrial fibrillation (irregular R-R intervals, absent P waves, fibrillatory waves), ventricular tachycardia (QRS >120 ms, rapid rate, often no discernible P waves), heart blocks (1st degree: PR interval >200 ms; 2nd degree: progressive PR prolongation until a QRS drops; 3rd degree: complete AV dissociation and atrial rate > ventricular rate) and premature contractions (early beats with wide or narrow QRS). Heart rate variability is analyzed via R-R interval variability over time (24-hour Holter), and the indicators include Time-Domain (SDNN and RMSSD) and Frequency-Domain (LF/HF ratio). Myocardial ischemia indicators include ST segment depression ≥0.5 mm in ≥2 contiguous leads, ST elevation ≥1 mm in ≥2 contiguous leads, and inversion or hyperacute T waves.
Cardiac evaluation by echocardiography | Within 3 days after enrollment
  Echocardiography data of all participants are acquired within 3 days after enrollment, in order to assess heart pumping function. Specifically, the key parameters assessed include ventricular function (ejection fraction: % of blood ejected per beat) and cardiac output quantification. The decline in the above indicators suggests heart ischemia or heart failure.
Cardiac evaluation by blood testing-1 | Within 3 days after enrollment
  Blood testing data of all participants are acquired within 3 days after enrollment and include several key cardiac biomarkers: myoglobin (normal: 14.3-65.8 μg/L), cardiac troponin I (cTnI, normal: 0-0.03 μg/L), cardiac troponin T (cTnT, normal: 0-0.1 μg/L), B-type natriuretic peptide (BNP, normal: 0-0.1 μg/L) and NT-proBNP (normal: <0.3 μg/L). Specifically, elevated myoglobin is useful for early detection of myocardial infarction (MI); elevated cTnI and cTnT, especially with a rising/falling pattern, are gold standard for diagnosing MI; elevated BNP and NT-proBNP suggest heart failure (HF), especially BNP >0.4 μg/L indicates severe HF.
Cardiac evaluation by blood testing-2 | Within 3 days after enrollment
  Blood testing data of all participants are acquired within 3 days after enrollment and include the following cardiac biomarkers: creatine kinase (CK, normal: 21-190 U/L ), CK-MB (normal: 0-25 U/L) and lactate dehydrogenase (LDH, normal: 114-240 U/L). Specifically, elevated CK and CK-MB suggest cardiac muscle injury; elevated LDH are useful for early detection of MI.

SECONDARY OUTCOMES:
Clinical prognosis assessed by GOS score | One month, three and six months after trauma
  Glasgow Outcome Scale (GOS) score (1 = death; 2 = persistent vegetative state; 3 = severe disability; 4 = moderate disability; 5 = good but not necessarily complete recovery; unfavorable outcome was defined as score of ≤3, and favorable outcome was defined as a score of >3)
Neurological function assessed by mRS score | One month, three and six months after trauma
  Modified Rankin Scale (mRS) score (0 = no symptoms; 1 = no significant disability; 2 = slight disability; 3 = moderate disability; 4 = moderately severe disability; 5 = severe disability; 6 = dead; favorable outcome was defined as score of 0-2, and unfavorable outcome was defined as score of 3-6)

CONTACTS AND LOCATIONS:
Overall Officials: Hao Chen, M.D., Ph.D., Study Director — Shanghai 6th Peoples' Hospital; Lai Wei, M.D., Principal Investigator — Shanghai 6th Peoples' Hospital
Locations (2):
- China (2):
  - Shanghai 6th People's Hospital, Shanghai
  - Shanghai Sixth People's Hospital, Shanghai